CLINICAL TRIAL: NCT01143389
Title: Evaluation of Two Riboflavin Dosing Regimens for Corneal Collagen Cross-Linking in Eyes With Progressive Keratoconus or Ectasia
Brief Title: Corneal Crosslinking in Patients With Keratoconus and Post-Refractive Ectasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-0243
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Keratoconus; Post-Refractive Ectasia
Keywords: Keratoconus; Ectasia; cross linking; collagen cross linking
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riboflavin 0.1% eyedrops every 5 minutes (Active Comparator): The eye will be irradiated for 30 minutes with UVX light, during which time instillation of riboflavin will continue (1 drop every 5 minutes for this arm).
  Interventions: Drug: Riboflavin; Device: UVX light
- Riboflavin 0.1% eyedrops every 2 minutes (Active Comparator): The eye will be irradiated for 30 minutes with UVX light, during which time instillation of riboflavin will continue (1 drop every 2 minutes for this arm).
  Interventions: Drug: Riboflavin; Device: UVX light

INTERVENTIONS:
Drug: Riboflavin — Riboflavin 0.1% eye drops are applied before and during irradiation of the cornea.
Device: UVX light — UVX 365 nm wavelength light source is applied with continued application of riboflavin.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using riboflavin and UV light to treat progressive keratoconus or post-refractive corneal ectasia.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate two riboflavin-dosing regimens for corneal collagen cross-linking to slow the progressive changes in corneal curvature in eyes with progressive keratoconus or post-refractive ectasia.

ELIGIBILITY:
Inclusion Criteria:

1. 10 years of age or older
2. Having documented ectasia on topography or tomography after previous refractive surgery OR progressive keratoconus defined as one or more of the following changes over a period of 36 months or less before randomization:

   1. An increase of ≥ 1.00 D in the steepest keratometry value (or sim K)
   2. An increase of ≥ 1.00 D in regular astigmatism evaluated by subjective manifest refraction
   3. A myopic shift (decrease in the spherical equivalent) of ≥ 0.50 D on subjective manifest refraction
   4. Documented decrease in visual acuity associated with irregular astigmatism and topographic features of ectasia.
3. Subjects with keratoconus diagnosis only:

   a. Axial topography consistent with keratoconus b. Presence of central or inferior steepening on the Pentacam map. c. Presence of one or more slit lamp findings associated with keratoconus, such as: i. Fleischer ring ii. Vogt striae iii. Corneal thinning iv. Corneal scarring
4. Contact Lens Wearers Only: Removal of contact lenses for the required period of time prior to the screening refraction:

   Contact Lens Type Minimum Discontinuation Time Soft 3 Days Soft Extended Wear 1 Week Soft Toric 2 Weeks Rigid gas permeable 2 Weeks
5. Signed written informed consent

Exclusion Criteria:

* 1. Any keratoconus patient over 21 years of age without evidence of progression of his corneal deformity.

  2. Patients with excessively thin corneas. 3. Previous ocular condition in the eyes to be treated that may predispose the eye for future complications, for example:

  a. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.) b. Clinically significant corneal scarring in the proposed treatment zone 4. A history of chemical injury or delayed epithelial healing in the eye(s) to be treated.

  5. A known sensitivity to treatment medications. 6. Patients with a current condition that, in the treating physician's opinion, would interfere with or prolong epithelial healing.

  7. Pregnancy (including plan to become pregnant) or lactation during the course of the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2010-05; Primary Completion 2017-05-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Wittig-Silva C, Whiting M, Lamoureux E, Lindsay RG, Sullivan LJ, Snibson GR. A randomized controlled trial of corneal collagen cross-linking in progressive keratoconus: preliminary results. J Refract Surg. 2008 Sep;24(7):S720-5. doi: 10.3928/1081597X-20080901-15. PMID 18811118
- [Background] Raiskup-Wolf F, Hoyer A, Spoerl E, Pillunat LE. Collagen crosslinking with riboflavin and ultraviolet-A light in keratoconus: long-term results. J Cataract Refract Surg. 2008 May;34(5):796-801. doi: 10.1016/j.jcrs.2007.12.039. PMID 18471635
- [Background] Mazzotta C, Traversi C, Baiocchi S, Sergio P, Caporossi T, Caporossi A. Conservative treatment of keratoconus by riboflavin-uva-induced cross-linking of corneal collagen: qualitative investigation. Eur J Ophthalmol. 2006 Jul-Aug;16(4):530-5. doi: 10.1177/112067210601600405. PMID 16952090
- [Background] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- [Derived] Price MO, Fairchild K, Feng MT, Price FW Jr. Prospective Randomized Trial of Corneal Cross-linking Riboflavin Dosing Frequencies for Treatment of Keratoconus and Corneal Ectasia. Ophthalmology. 2018 Apr;125(4):505-511. doi: 10.1016/j.ophtha.2017.10.034. Epub 2017 Dec 2. PMID 29203068
- See also: Price Vision Group Website — http://www.pricevisiongroup.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Riboflavin 0.1% Eyedrops Every 5 Minutes: The eye will be irradiated for 30 minutes with UVX light, during which the instillation of riboflavin will continue (1 drop every 5 minutes for this arm).
  Riboflavin: Riboflavin 0.1% eye drops are applied before and during irradiation of the cornea.
  UVX light: UVX 365 nm wavelength light source is applied with continued application of riboflavin.
- Riboflavin 0.1% Eyedrops Every 2 Minutes: The eye will be irradiated for 30 minutes with UVX light, during which the instillation of riboflavin will continue (1 drop every 2 minutes for this arm).
  Riboflavin: Riboflavin 0.1% eye drops are applied before and during irradiation of the cornea.
  UVX light: UVX 365 nm wavelength light source is applied with continued application of riboflavin.
Period: Overall Study
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
Started | 253 | 257
Completed | 227 | 232
Not Completed | 26 | 25
Not completed — Lost to Follow-up | 26 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes | Total
Number analyzed (Participants) | 253 | 257 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (12) | 32 (13) | 32 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 191 | 196 | 387
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 13 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 24 | 52
  White | 215 | 220 | 435
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 253 | 257 | 510
Keratoconus/ectasia classification [Count of Participants; unit: Participants] — Patients with keratoconus were classified as mild, moderate, or severe based upon tomography imaging of the shape of the anterior corneal surface. The imaging device reports the keratometry (curvature) in the steep meridian and the orthogonal flat meridian. The keratoconus was classified as mild if the flat keratometry was less than 51 diopters. Keratoconus was classified as moderate if the flat keratometry was between 51 and 56 diopters or astigmatism exceeded 8 diopters. Keratoconus was classified as severe if the flat keratometry exceeded 56 diopters.
  Participants
    Keratoconus mild (flat K <51D and astigmatism <8D) | 140 | 139 | 279
    Keratoconus moderate | 43 | 43 | 86
    Keratoconus severe (flat K >56D by tomography) | 20 | 21 | 41
    Ectasia after refractive surgery | 50 | 54 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Keratometry From Baseline to 6 Months After Treatment
Description: Change in maximum keratometry (Kmax) between baseline and 6 months after treatment, measured by corneal tomography.
Time Frame: 6 months
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
Number analyzed (Participants) | 227 | 232
diopters | 0.76 (2.4) | 0.97 (3.2)

2. Secondary Outcome: Pachymetry
Description: Minimum corneal thickness measured by corneal tomography
Time Frame: 6 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
Number analyzed (Participants) | 227 | 232
microns | 438 (51) | 434 (20)

3. Secondary Outcome: Corrected Distance Visual Acuity (CDVA)
Description: Corrected distance visual acuity (CDVA) reported in logarithm of the minimum angle of resolution (logMAR). Lower numbers represent better vision; 0.0 corresponds to 20/20 vision. Each increase of 0.1 on the logMAR scale corresponds to one less line read on the eye chart.
Time Frame: 6 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
Number analyzed (Participants) | 227 | 232
logMAR | 0.32 (0.29) | 0.31 (0.28)

4. Secondary Outcome: Uncorrected Distance Visual Acuity (UDVA)
Description: Uncorrected distance visual acuity reported in logarithm of the minimum angle of resolution units. Lower numbers represent better vision; 0.0 corresponds to 20/20 vision without any type of correction such as glasses. Each increase of 0.1 on the logMAR scale corresponds to one less line read on the eye chart.
Time Frame: 6 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
Number analyzed (Participants) | 227 | 232
logMAR | 0.95 (0.53) | 0.91 (0.55)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Riboflavin 0.1% Eyedrops Every 5 Minutes | Riboflavin 0.1% Eyedrops Every 2 Minutes
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/257
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/257
Other Adverse Events (participants affected / at risk) | 12/253 | 13/257
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riboflavin 0.1% Eyedrops Every 5 Minutes (N=253) | Riboflavin 0.1% Eyedrops Every 2 Minutes (N=257)
Loss of 2 or more logMAR lines of corrected distance visual acuity (CDVA) relative to baseline (Eye disorders) | 12 (12) | 13 (13)

LIMITATIONS AND CAVEATS:
Limitations included the 6-month follow up duration and the reduced reproducibility of measurement techniques in eyes with ectasia as compared with normal eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT01143389/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT01143389/SAP_002.pdf